CLINICAL TRIAL: NCT00976092
Title: Randomized Trial of Prasugrel Plus Bivalirudin vs. Clopidogrel Plus Heparin in Patients With Acute STEMI
Brief Title: Efficacy Study of Combined Prasugrel and Bivalirudin Versus Clopidogrel and Heparin in Myocardial Infarction
Acronym: BRAVE-4
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE I01209
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; clopidogrel; prasugrel; bivalirudin; primary PCI
MeSH Terms: conditions — Myocardial Infarction | interventions — Prasugrel Hydrochloride; bivalirudin; Clopidogrel; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel + Bivalirudin (Experimental): 60 mg prasugrel plus bivalirudin
  Interventions: Drug: Prasugrel; Drug: Bivalirudin
- Clopidogrel + Heparin (Active Comparator): clopidogrel as loading and heparin
  Interventions: Drug: Clopidogrel; Drug: Heparin

INTERVENTIONS:
Drug: Prasugrel — 60 mg prasugrel as loading dose prior to PPCI
  Other Names: Efient
  Arms: Prasugrel + Bivalirudin
Drug: Bivalirudin — IV bolus 0.75 mg/kg of body weight followed by an infusion of 1.75 mg/kg/hour during the PPCI
  Other Names: Angiox
  Arms: Prasugrel + Bivalirudin
Drug: Clopidogrel — 600 mg clopidogrel as loading dose before PPCI
  Other Names: Plavix
  Arms: Clopidogrel + Heparin
Drug: Heparin — i.v. bolus of 70-100 IU/kg body weight
  Other Names: unfractionated Heparin
  Arms: Clopidogrel + Heparin

SUMMARY:
Randomized comparison of two different anticoagulation strategies: prasugrel plus bivalirudin versus clopidogrel plus heparin in patients with acute myocardial infarction undergoing emergency catheterization and coronary intervention.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PPCI) is the preferred reperfusion strategy for patients with acute ST-segment elevation myocardial infarction (STEMI). Additional anticoagulation therapy prior or during intervention plays an important role in the short- and long-term outcomes after PPCI. Two separate studies have shown significant benefit against conventional therapy based on clopidogrel and heparin for two recently approved drugs: the direct thrombin inhibitor bivalirudin and the thienopyridine prasugrel. In the HORIZONS-AMI trial, bivalirudin after pretreatment with clopidogrel resulted in improved net clinical outcomes. However, during the first 24 hours after PPCI an increase in the stent thrombosis rate was observed with bivalirudin therapy. Prasugrel has been shown to be superior to clopidogrel in patients with acute coronary syndromes undergoing PCI. The benefit in reduction of ischemic complication was even greater in the subset of patients with STEMI without any increase in the bleeding risk and with a significant reduction in the stent thrombosis rate. Expectedly, the synergic actions of prasugrel and bivalirudin may maximize the benefit of antithrombotic therapy for STEMI patients undergoing PPCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting within 24 hours from the onset of symptoms with STEMI
2. Informed, written consent
3. In women with childbearing potential a pregnancy test is obligatory.

Exclusion Criteria:

1. Age < 18 years
2. Cardiogenic shock
3. Active bleeding; bleeding diathesis; coagulopathy
4. History of gastrointestinal or genitourinary bleeding <2 months
5. Refusal to receive blood transfusion
6. Major surgery in the last 6 weeks
7. History of intracranial bleeding or structural abnormalities
8. Suspected aortic dissection
9. Heparin-induced thrombocytopenia
10. Any previous stroke
11. Prior administration of thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux for the index MI
12. Known relevant hematological deviations: Hb <100g/l, Thromb. <100x10^9/l
13. Use of coumadin derivatives within the last 7 days
14. Chronic therapy with nonsteroidal anti-inflammatory drugs (except aspirin), COX-2 inhibitors, prasugrel
15. Known malignancies or other comorbid conditions with life expectancy <1 year
16. Known severe liver disease, severe renal failure
17. Known allergy to the study medications
18. Previous enrollment in this trial
19. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
composite of all-cause death, recurrent MI, unplanned IRA revascularization, stroke, definite stent thrombosis or major bleeding | 30 days

SECONDARY OUTCOMES:
all-cause death, recurrent MI, unplanned IRA-revascularization, stroke or definite stent thrombosis | 30 days
major bleeding complications | 30 days
cardiac death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (3):
- Germany (3):
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Klinikum rechts der Isar, Technische Universitaet Muenchen, Munich, Bavaria
  - Herzzentrum der Segeberger Kliniken, Bad Segeberg

REFERENCES:
- [Derived] Schulz S, Richardt G, Laugwitz KL, Morath T, Neudecker J, Hoppmann P, Mehran R, Gershlick AH, Tolg R, Anette Fiedler K, Abdel-Wahab M, Kufner S, Schneider S, Schunkert H, Ibrahim T, Mehilli J, Kastrati A; Bavarian Reperfusion Alternatives Evaluation (BRAVE) 4 Investigators. Prasugrel plus bivalirudin vs. clopidogrel plus heparin in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2014 Sep 7;35(34):2285-94. doi: 10.1093/eurheartj/ehu182. Epub 2014 May 9. PMID 24816809
- [Derived] Schulz S, Richardt G, Laugwitz KL, Mehran R, Gershlick AH, Morath T, Mayer K, Neudecker J, Tolg R, Ibrahim T, Hauschke D, Braun D, Schunkert H, Kastrati A, Mehilli J; Bavarian Reperfusion Alternatives Evaluation (BRAVE) 4 Investigators. Comparison of prasugrel and bivalirudin vs clopidogrel and heparin in patients with ST-segment elevation myocardial infarction: Design and rationale of the Bavarian Reperfusion Alternatives Evaluation (BRAVE) 4 trial. Clin Cardiol. 2014 May;37(5):270-6. doi: 10.1002/clc.22268. Epub 2014 Mar 14. PMID 24633823